CLINICAL TRIAL: NCT06118346
Title: A Female-Specific Cognitive Behavioral Therapy Group for Alcohol Use Disorder in VA Primary Care Settings
Brief Title: A Female-Specific CBT Group for Veteran Women With Alcohol Use Disorder in VA Primary Care Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Epstein, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H00021304; 1R01AA028240-01A1 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-11-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Risky Health Behavior
MeSH Terms: conditions — Alcoholism; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Female-Specific Cognitive Behavioral Therapy (Experimental): Participants in this arm will receive female-specific cognitive behavioral therapy and usual VA care for alcohol use disorder.
  Interventions: Behavioral: Female-Specific Cognitive Behavioral Therapy (FS-CBT); Behavioral: Usual Care
- Usual Care (Active Comparator): Participants in this arm will receive usual VA care for alcohol use disorder.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Female-Specific Cognitive Behavioral Therapy (FS-CBT) — FS-CBT is a unique 12-session weekly group CBT treatment designed for women Veterans with AUD and/or risky drinking, and provides (1) AUD interventions, (2) general female-specific content, (3) female-Veteran content, (4) wellness and self-care, and (5) a novel 24/7 social support for abstinence discussion mobile app.
  Arms: Female-Specific Cognitive Behavioral Therapy
Behavioral: Usual Care — Usual care means that participants will receive brief alcohol counseling and have access to available treatments for AUD at the VA.

SUMMARY:
The purpose of this study is to evaluate a Female-Specific Cognitive Behavioral Therapy (CBT) Group as treatment for Alcohol Use Disorder among Veteran women.

DETAILED DESCRIPTION:
This is a five year Hybrid Type 1 effectiveness-implementation study. For Aim 1, 162 female Veterans with AUD will be enrolled over 2.5 years in the study at Primary Care and Women's Comprehensive Primary Care Clinics (i.e., the Women's Health Clinic) in the VA New York Harbor Healthcare System (VA NYHHS) (n=162) for a final sample of 140 at 15 month post-baseline (i.e.,12 month post treatment) follow up. The 86% follow up rate is based on Dr. Epstein's prior Randomized Control Trial (RCT) testing FS-CBT for civilian women with AUD on which the current Veteran- Centric FS-CBT group is based. After the research baseline interview, participants will be randomly assigned to either Usual Care (UC, which is Brief Alcohol Counseling +Referral to Substance Use Disorder (SUD) Specialty Care if indicated, all called Brief Alcohol Counselling (BAC), and otherwise also known as Brief Intervention and Referral to treatment (BIRT)) or to the 12 session, rolling entry group Veteran Female Specific CBT for AUD (FS-CBT) held within the VA NYHHS Women's Health Clinic. Participants in both conditions will complete the same baseline (BL), 3-, 9- and 15-months post-BL (i.e., 0-, 6-, & 12-months after treatment) research assessments. Primary outcome variables will be treatment access (attending least one FS- CBT group session or 1 SUD specialty care session in the FS-CBT condition, and at least 1 SUD specialty care session in the usual UC condition; treatment engagement is defined as number of treatment hours attended in each condition); drinking outcomes (percent drinking days and percent heavy drinking days during and 1 year after the treatment phase). Secondary outcomes include drug use, mental health, social support for abstinence, and health behaviors. For Aim 2, a formative evaluation will be done during the RCT using program process data to track provider interest, patient enrollment rates, reasons for refusal, and treatment adherence.

Using an implementation science framework (Consolidated Framework for Implementation Research, CFIR), the investigators will evaluate implementation barriers and facilitators of FS-CBT in VA PC using qualitative interviews with 20 women Veterans in FS-CBT, 20 in UC, 15 women with AUD who were eligible but did not enroll in the RCT, and 16 providers/stakeholders. The goal of the formative evaluation is to help determine factors at the system, provider, and patient levels that affect the likelihood that FS-CBT will be successfully implemented and sustained in VA Primary Care (PC). The evaluation will allow for more rapid translational gains in terms of intervention uptake and sustainability. The evaluation will include the systematic collection of quantitative RCT process data (e.g., number and % of patient referral opt-outs by Primary Care Providers (PCPs), % of eligible women who enroll, reasons for refusal, number of group sessions completed by Veteran characteristics), and qualitative data via interviews with patient and staff stakeholders. To learn about patient-level barriers/facilitators, study personnel will conduct interviews with 20 female Veterans who were randomized to the FS-CBT condition, and 20 who were randomized to UC: (a) one-half will be drawn from those who completed the full dose (12 sessions in FS-CBT and all treatment recommendations in UC) and the other half from those who dropped out and completed less than the recommended minimal dose. Investigators will sample from participants who significantly reduced their drinking and from those who did not. Investigators will include a diverse sample of Veterans based on age, gender, race/ethnicity, era of military service, and diagnoses (e.g., PTSD). Lastly, study personnel will interview 15 women with AUD who were eligible but did not enroll in the RCT to understand their perceptions of the program and barriers to participation.

The CFIR framework will be used to guide the interview approach. CFIR is a typology of 39 constructs from five main domains that identify factors associated with successful implementation and maintenance of health care innovations: (1) Intervention Characteristics; (2) Inner Setting; (3) Outer Setting; Characteristics of Individuals; (5) Process. If Aim 1 hypotheses are supported, these interviews will help guide subsequent implementation trials of FS-CBT by explaining: (a) barriers and facilitators to participation; perceptions about why FS-CBT is successful at achieving better outcomes for women Veterans with AUD; the barriers and facilitators to high fidelity implementation of FS-CBT; and the sustainability of FS-CBT in the absence of a funded research project and how to achieve this goal; and (b) how FS-CBT should be adjusted to appeal to the subgroup of Veterans. If Aim 1 hypotheses are not supported, the interviews will determine the reasons why (i.e., questions posed to staff and patients will solicit information on barriers associated with delivery of FS-CBT during the RCT, and what modifications to FS-CBT could be made to maximize effectiveness).

ELIGIBILITY:
Inclusion criteria:

* women aged 18 or older
* Veteran of the U.S. Armed Forces
* Enrolled in healthcare at VA NYHHS;
* AUDIT-C ≥3 plus diagnosis of AUD and/or risky drinking (defined by the National Institute on Alcohol Abuse and Alcoholism as more than 3 drinks on any one day or more than 7 drinks per week) on more detailed screening
* consumed alcohol within 90 days prior to our study's initial eligibility screen.

Exclusion criteria:

* participant is acutely suicidal
* participant has acute psychotic or manic symptoms associated with severe mental illness
* participant is pregnant at initial eligibility screen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — identifies as a woman
Enrollment: 162 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems
Structured Clinical Interview for DSM Disorders (SCID) Alcohol Use Disorder Module | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  semi-structured interview that assesses for alcohol use disorder based on the Diagnostic and Statistical Manual for Mental Disorders (DSM)
Form 90 Timeline Followback (TLFB) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  interview used to assess alcohol and drug use over a specific period of time
Treatment Services Review (TSR) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  interview used to assess use of Veterans Affairs and non-Veterans Affairs treatments including Alcohol Use Disorder treatment, physical and mental health treatment, and use of medications
Electronic Medical Record (EMR) | assessed from baseline to 15-months post-baseline follow-up
  patient's medical records - review to assess use of Veterans Affairs and non-Veterans Affairs treatments including Alcohol Use Disorder treatment, physical and mental health treatment, and use of medications

SECONDARY OUTCOMES:
Outcome Questionnaire-45 | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  self-report questionnaire used to rate symptoms, interpersonal problems, and social role dysfunction
Posttraumatic Stress Disorder Checklist (PCL)-5 with Life Events Checklist (LEC)-5 | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  combined self-report questionnaire and interview used to measure posttraumatic stress disorder symptoms
Difficulties in Emotion Regulation Scale (DERS) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  self-report questionnaire that assesses emotion regulation
Coping Strategies Scale (CSS) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  self-report questionnaire used to assess use of coping strategies
Important People Interview (IPI) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  interview used to assess social network characteristics
Sociotropy Autonomy Scale (SAS) | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  self-report questionnaire used to assess the two personality dimensions of sociotropy and autonomy
Use of Women2Women mobile application | assessed from baseline to 15-months post-baseline follow-up
  tracking use of mobile app designed to allow participants randomized to the FS-CBT (female-specific cognitive behavioral therapy) + UC (usual care) to interact with and provide support to one another
Self-Care Questionnaire | assessed at baseline, and 3-, 9-, and 15-months post-baseline follow-up
  self-report questionnaire used to assess level of self-care

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Epstein, PHD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No